CLINICAL TRIAL: NCT05290311
Title: What Are the Long-Term Effects of Cognitive-Behavioural Therapy on Quality of Life in Adult Patients With ADHD?
Brief Title: Long-Term Effects of CBT on Quality of Life in Adults With ADHD
Acronym: CBT-QoL
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, R.K.R.W. Wettstein, Research Coordinator, Amsterdam UMC, location VUmc
Other Study IDs: NL79674.018.22
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: cognitive behavioural therapy; CBT; ADHD; self-esteem; self-efficacy; Rosenberg Self-Esteem Scale; Generalized Self-Efficacy Scale; long term outcomes; ADHD-RS-IV scale; AAQoL scale; socio-economic status; SES; income; occupation; housing situation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COMB: The 'combined' or 'COMB' group received cognitive behavioural therapy next to pharmacotherapy for ADHD in the past. Patients chose themselves whether or not they wanted to receive cognitive behavioural therapy.
  Interventions: Behavioral: cognitive behavioural therapy
- PHA: The 'pharmacotherapy' group or 'PHA' received pharmacotherapy for ADHD only in the past. Patients chose themselves whether or not they wanted to receive cognitive behavioural therapy.

INTERVENTIONS:
Behavioral: cognitive behavioural therapy — Cognitive behavioural therapy (CBT) was given according to the protocol of Safren (2004, 2005). Each participant followed one session of 60 minutes per week, for 10 to 16 weeks. Psychotherapists giving CBT had at least a master diploma.
  Other Names: Pharmacotherapy
  Groups: COMB

SUMMARY:
Background and objective: Although the short-term effects of cognitive behavioural therapy (CBT) in adult patients with ADHD are established, not a lot is known about longer-term effects. To assess the additive value of CBT to pharmacotherapy in the long term, an assessment of ADHD symptoms and quality of life in patients that followed CBT four to eight years ago is done. To understand how CBT impacts quality of life in patients, an assessment of self-efficacy and self-esteem is made. Furthermore, patients will be asked whether they currently still use medicine for ADHD and CBT strategies. To evaluate whether CBT impacts the economic situation of the patient, an assessment of income, occupation status and the housing situation of the patient is done.

Study Design: As this is a follow-up, observational cohort study, the same patients from Wettstein et al. (2021) are invited for participation. During February and March, patients are informed via email about the study. Online, patients are asked to provide informed consent and are able to fill in the complete questionnaire. The duration of the questionnaire is 45 minutes and each patient is compensated with a 25 Euro gift card.

Outcome variables: ADHD symptoms are measured on the ADHD-RS-IV, quality of life is measured on the AAQoL scale, self-efficacy is measured on the GSES, and self-esteem is measured on the RSES. Medication status, CBT strategy use and data about the socioeconomic status of the patient is asked in multiple choice questions.

DETAILED DESCRIPTION:
Background of the study:

Cognitive behavioral therapy (CBT) in adult patients with ADHD teaches the patient strategies to compensate for the problems their symptoms produce in daily life. Next to this, CBT achieves to challenge the negative cognitions which patients with ADHD have developed because of their symptoms during lifetime. Research during the previous years has shown that CBT is effective in reducing ADHD symptoms in adult patients. Little research is done about the effects of CBT on quality of life (QoL). The largest study so far assessing QoL in adult patients with ADHD is conducted by Wettstein et al. (2021). The authors compared patients that received CBT next to pharmacotherapy with patients that received pharmacotherapy only on the Adult ADHD Quality of Life (AAQoL) scale. No difference has been found between both groups post-treatment. As CBT teaches strategies that have to be learned and trained over time, it is likely that also effects on QoL might require time to develop. Support for this theory has been found by Cherkasova et al. (2020) that compared CBT-alone with CBT in combination with pharmacotherapy in adult patients with ADHD. While the CBT-only condition scored significantly lower on ADHD-symptom ratings compared to the combination group, these differences became smaller and even insignificant after six months. Other publications report a similar effect for measures of self-esteem and self-efficacy after CBT for ADHD in adults.

Primary Objective:

To identify whether CBT in combination with pharmacotherapy improves the quality of life in adult patients with ADHD four to eight years after treatment. To identify if CBT in addition to pharmacotherapy is associated with increased medication use and by this, symptom control, over time. An attempt is done to understand how CBT works in the long term by measuring self-esteem and self-efficacy in patients that did or did not chose for CBT treatment. To understand the impact of CBT treatment on the economic position of the patient, an estimate of the socioeconomic status will be assessed.

Study Design:

The study will be a observational, follow-up, cohort study. The study will be a follow-up of Wettstein et al. (2021) and is supposed to take place during May to June 2022 at the AMC (Amsterdam Medical Center) hospital. Patient data of five different GGZ (Geestelijke Gezondheidszorg) centra in the Netherlands specialized in the treatment of ADHD in adults will be collected (ADHDcentraal: Utrecht, Amsterdam, Rotterdam, Nijmegen, Zwolle). Data will be analyzed and an article will be written and published during July to December 2022.

Quality assurance plan:

This study is registered at the METC AMC, Amsterdam. Data monitoring is conducted by the Clinical research Monitoring Center, AMC hospital. Prior to study registration, a risk assessment analysis has been done according to AMC hospital guidelines. This study is recorded under clinicaltrials.gov before registration.

All documents delivered to the patients are pre-designed. To ensure safety of data assessment, all data will be collected online via the clinical trial platform Castor EPD.

Primary study parameters/outcome of the study:

Only well-researched neuropsychological instruments are used. Quality of life, measured on the Adult ADHD Quality of Life (AAQoL) scale Description: The AAQoL Scale consists out of 29 items and asks the patient how often he/she experienced a given situation. Each item is rated on a 5-point Likert scale. The scale consists out of four subscales (productivity, life outlook, relationships, psychological health)which are confirmed by factor analysis.

Description: The ADHD-RS-IV scale consists out of 18 items that are rated on a 4-point Likert scale. The frequency of ADHD-related symptoms during the previous 6 months is assessed. There are two subscales (inattention and hyperactive-impulsive) that are related to the two symptom dimensions of ADHD described in the DSM-IV.

Self-efficacy, measured on the General Self-Efficacy Scale (GSES) Description: The GSES scale consists out of 10-items which are rated on a 4-point Likert scale. The scale measures the concept of generalized self-efficacy, "characterized by a broad and stable sense of personal competence about coping effectively with diverse stressful situations".

Self-esteem, measured on the Rosenberg Self-Esteem Scale (RSES) The RSES consists out of 10 items rated on a 4-point Likert scale. The scale assesses global self-esteem, measuring "a favorable or unfavorable attitude towards the self".

Socioeconomic status (SES) Two questions are asked about the SES of the patient. One question asks about the monthly brutto income. A second question asks about the occupation of the patient and provides four options to answer (full-time/part-time/no occupation/I would rather not like to tell). One question will be asked about the housing situation of the patient with multiple choice answer options (own house, own apartment, rented house, rented apartment, in a shared flat) Use of medication The following question will be asked: Do you still use medication for ADHD?. Two answer options are provided (Yes/No).

Use of CBT strategies One question is asked about whether the patient still uses strategies learned during CBT. In a multiple-choice question, 13 different strategies are possible to select.

Data about the socio-economic status of the patient will be compared to Dutch national comparison data from the year 2022.

Procedure:

All patients that participated in Wettstein et al. (2021) and gave consent to be informed about future studies are invited for study participation in May 2022. Via Email, each patient is informed about the current study. Via a link, each patient is asked to provide informed consent. After giving consent, the patient can procede to the online questionnaire. The duration of the complete questionnaire is approximately 45 minutes.

Sample size assessment:

The same population included in Wettstein et al. (2021) will be invited for participation. All subjects were drawn from the patient population of a Dutch mental health care provider.

Statistical Analysis Plan:

Descriptive statistics will be requested for all outcome variables as well as the characteristics of the sample (gender, age, location at which patient was treated).

AAQoL, ADHD-RS-IV, GSES, RSES scores and income data will be compared for both groups (CBT vs. no CBT) in an ANOVA model. The assumptions of the ANOVA model will be tested prior to analysis. When a significant effect is found, pairwise comparisons are done with a Bonferroni correction. The following calculations will be reported: Mean and standard deviation, F-value, t-value, 95% confidence interval, degrees of freedom, p-value and effect size Medication status, CBT strategy use, and housing data and occupation data are analyzed in a chi-square model. The assumptions of the chi-square model will be evaluated prior to analysis. The following calculations will be reported: Mean and standard deviation, Pearson's Chi-Square, 95% confidence interval, degrees of freedom, p-value and effect size.

Data on income, occupation status and housing will be compared to the national average.

Missing data will be addressed in a best case/worst case analysis. Data analysis will be supported by a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the study by Wettstein et al. (2021).

Exclusion Criteria:

* Not applicable as this is a follow-up study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The gender distribution in the sample is approximately 1:1. All participants should be aged between 18 and 70 years. The estimation is based according to the original sample distribution.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Quality of life, measured with the Adult ADHD Quality of life scale (AAQoL) | 5 to 10 minutes
  Quality of life is measured with the Adult ADHD Quality of life (AAQoL) Scale. Outcome is the mean change in total score from baseline and post-treatment to follow-up assessment. To calculate the total score, the domainscores of the subscales life productivity, relationships and psychological health are turned around. All scores are transverted to a scale of 100 (1 = 0, 2 = 25, 3 = 50, 4 = 75, 5 = 100). All scores are summed up and divided by the amount of items. The maximum score ranges from 0 to 100, with higher scores indicating a better life quality.
ADHD Symptoms, measured with the ADHD-RS-IV scale | 5 to 10 minutes
  ADHD Symptoms are measured with the ADHD Rating Scale IV (ADHD-RS-IV). Outcome is the mean change in total score from baseline and post-treatment to follow-up assessment per group. Total scores range from 0 to 54, higher scores indicating more symptoms.
Self-Esteem, measured with the Rosenberg Self-Esteem Scale (RSES) | 5 minutes
  Self-Esteem is measured with the Rosenberg Self-Esteem Scale. Outcome is the mean total score on the scale per group. Total scores range from 0 to 30 points, with higher scores indicating a higher self-esteem.
Self-Efficacy, measured with the Generalized Self-Efficacy Scale (GSES) | 5 minutes
  Self-Efficacy is measured with the Generalized Self-Efficacy Scale. Outcome is the mean total score on the scale per group. Total scores range from 10 to 40 points, higher scores indicate high self-efficacy.
Medication status, measured with a multiple-choice question | < 5 minutes
  Medication status of the patient is measured with one multiple choice question. Outcome is the total number of participants currently using medication per group.
CBT strategy use, measured with a multiple-choice question | 5 minutes
  Use of CBT strategies is measured by one multiple choice question. Outcome is the total number of participants currently using each strategy, as well as the average number of strategies used per group.
Socioeconomic status | 5 minutes
  Socioeconomic status is measured by three open or multiple choice questions, one regarding income, one regarding occupation status and one regarding the housing situation of the patient. Outcome is the average income and the average distribution of the sample in occupation status and housing situation per group.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Dumont, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- ADHDcentraal, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wettstein RKRW, Klabbers Y, Romijn E, Nieuwveen J, Kroesen JC, Wettstein KRM, Dumont GJH. [Cognitive behavioral therapy in combination with pharmacotherapy for adults with ADHD]. Tijdschr Psychiatr. 2021;63(7):550-556. Dutch. PMID 34523707